CLINICAL TRIAL: NCT01673594
Title: Prevention of Stimulant-Induced Euphoria With an Opioid Receptor Antagonist
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Thomas J. Spencer, MD, Associate Chief, Clinical and Research Program, Pediatric Psychopharmacology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-P-000918
Record Dates: First submitted 2012-06-21; First posted 2012-08-28 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: ADHD; Stimulant-Induced Euphoria
Keywords: ADHD; Naltrexone; SODAS MPH; Stimulant-Induced Euphoria; Substance Abuse; Adults
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Substance-Related Disorders | interventions — Methylphenidate; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone (Experimental): Arm 1: Naltrexone + SODAS MPH
  Interventions: Drug: SODAS MPH; Drug: Naltrexone
- Placebo (Placebo Comparator): Arm 2: Placebo + SODAS MPH
  Interventions: Drug: SODAS MPH

INTERVENTIONS:
Drug: SODAS MPH — Adults with ADHD will receive open-label SODAS MPH
  Other Names: Ritalin LA
Drug: Naltrexone — Subjects randomized to the "active" double-blind group will receive Naltrexone HCl
  Other Names: Naltrexone HCl
  Arms: Naltrexone

SUMMARY:
The purpose of this study is to a) assess the efficacy of naltrexone in preventing stimulant-induced euphoria in adults with ADHD, b) assess whether naltrexone will interfere with the clinical efficacy of stimulants in treating adults with ADHD, c) assess whether naltrexone will interfere with the effects of stimulants on neurotransmitter activity. We predict that naltrexone will successfully prevent stimulant-induced euphoria without interfering with the ability of stimulants to effectively treat ADHD in adults. This study will be an 8 -week trial with young adults (18-24) with ADHD.

ELIGIBILITY:
Inclusion

1. Male and female outpatients
2. age 18-30
3. diagnosis of ADHD by DSM-IV, per clinical evaluation and confirmed by structured interview
4. likeability response (> 5) on Question #2 of the DRQ-S after an initial test dose of 60 mg of IR MPH.
5. Baseline ADHD severity of > 20 on the Adult ADHD Investigator System Report Scale (AISRS)
6. Able to participate in blood draws and to swallow pills.
7. Subjects must be considered reliable reporters, must understand the nature of the study and must sign an informed consent document

Exclusion

1. Any current (last month), non-ADHD Axis I psychiatric conditions
2. Ham-D > 16, BDI > 19, or Ham-A > 21
3. Any clinically significant chronic medical condition
4. any cardiovascular disease or hypertension
5. Clinically significant abnormal baseline laboratory values
6. I.Q. < 80)
7. Organic brain disorders
8. Seizures or tics
9. Pregnant or nursing females
10. Clinically unstable psychiatric conditions (i.e. suicidal behaviors, psychosis)
11. Current or recent (within the past year) substance abuse/dependence
12. patients on other psychotropics
13. Current or prior adequate treatment with MPH
14. known hypersensitivity to methylphenidate
15. Current opioid use (by history and urine screen) or potential need for opioid analgesics during the study
16. acute hepatitis or liver failure (baseline blood tests).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Spencer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Spencer TJ, Bhide P, Zhu J, Faraone SV, Fitzgerald M, Yule AM, Uchida M, Spencer AE, Hall AM, Koster AJ, Feinberg L, Kassabian S, Storch B, Biederman J. The Mixed Opioid Receptor Antagonist Naltrexone Mitigates Stimulant-Induced Euphoria: A Double-Blind, Placebo-Controlled Trial of Naltrexone. J Clin Psychiatry. 2018 Mar/Apr;79(2):17m11609. doi: 10.4088/JCP.17m11609. PMID 29617066
- [Derived] Spencer TJ, Bhide P, Zhu J, Faraone SV, Fitzgerald M, Yule AM, Uchida M, Spencer AE, Hall AM, Koster AJ, Biederman J. Opiate Antagonists Do Not Interfere With the Clinical Benefits of Stimulants in ADHD: A Double-Blind, Placebo-Controlled Trial of the Mixed Opioid Receptor Antagonist Naltrexone. J Clin Psychiatry. 2018 Jan/Feb;79(1):16m11012. doi: 10.4088/JCP.16m11012. PMID 28640990

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naltrexone | Placebo
Started | 18 | 19
Completed | 12 | 13
Not Completed | 6 | 6
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 2 | 4
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for subjects who made it to week 3 of the trial and were included in analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.1 (2.9) | 24.4 (3.2) | 24.8 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 10 | 13 | 23
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Score on AISRS From Baseline to Week 6
Description: The Adult ADHD Investigator System Report Scale (AISRS) is an 18-item, DSM-IV symptom Likert scale that measures ADHD symptoms in adults. Each of the individual symptoms of ADHD is rated from 0 to 3 on a scale of severity (3 being more severe symptoms). Total scores range from 0 to 54; higher scores indicate greater symptom severity. Change was calculated as value at baseline minus value at 6 weeks.
Time Frame: Baseline and 6 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 12 | 13
units on a scale | -26.7 (10.1) | -29.1 (10.0)

2. Primary Outcome: Safety
Description: Number of adverse events throughout the course of the study
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: adverse events
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 15 | 16
adverse events | 6.73 (4.7) | 4.75 (3.4)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 18/18 | 16/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone (N=18) | Placebo (N=19)
Cold/Infection/Allergy (General disorders) | 2 (2) | 4 (5)
Decreased appetite (Metabolism and nutrition disorders) | 5 (13) | 1 (2)
Headache (Nervous system disorders) | 8 (20) | 7 (16)
Nausea/Vomit/Diarrhea (Gastrointestinal disorders) | 12 (19) | 8 (9)
Insomnia (Nervous system disorders) | 8 (14) | 7 (13)
Sedation (Nervous system disorders) | 0 (0) | 1 (1)
Decreased Energy (Psychiatric disorders) | 4 (4) | 1 (1)
Increased Energy (Psychiatric disorders) | 2 (2) | 0 (0)
Cardiovascular (Cardiac disorders) | 1 (1) | 4 (5)
Tense/Jittery (Psychiatric disorders) | 5 (7) | 3 (5)
Agitated/irritable (Psychiatric disorders) | 4 (4) | 0 (0)
Sad/Down (Psychiatric disorders) | 3 (5) | 2 (2)
Anxious/Worried (Psychiatric disorders) | 1 (1) | 3 (3)
Autonomic: Drool/Sweat (General disorders) | 2 (2) | 2 (3)
Mucosal Dryness (General disorders) | 2 (4) | 1 (1)
DizzyLightheaded (Nervous system disorders) | 0 (0) | 1 (1)
Extra Pyramidal Symptoms (Nervous system disorders) | 0 (0) | 1 (1)
Neurological (Nervous system disorders) | 1 (1) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (5)
Dermatological (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pressure (General disorders) | 1 (1) | 0 (0)
Feels Warm (General disorders) | 1 (2) | 0 (0)
Unable to Feel Emotions (Psychiatric disorders) | 0 (0) | 1 (1)
Tingly Feeling in Head and Chest (General disorders) | 0 (0) | 1 (1)
Menstrual Cramps (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No